CLINICAL TRIAL: NCT01942499
Title: A Randomized Controlled Trial of a Post-rehabilitation Community-based Exercise Program for Individuals With COPD
Brief Title: Community-Based Maintenance Exercise Program for COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Collaborators: Ontario Lung Association (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Roger Goldstein, Respirologist, West Park Healthcare Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-006-WP
Record Dates: First submitted 2013-09-04; First posted 2013-09-16 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, exercise, community
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Exercise Group (Other): Community-based exercise program for one year
  Interventions: Other: Community-based exercise program
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Community-based exercise program
  Arms: Community Exercise Group

SUMMARY:
It is well established that individuals living with chronic obstructive pulmonary disease (COPD) demonstrate significant improvements following a formal rehabilitation program. The problem lies in the fact that these functional improvements diminish over a 12 month period. This decline in function is associated with decreased participation, a decline in health status, and an increased need to access the healthcare system. The objective of this project is to evaluate the effectiveness of a post-rehabilitation community-based exercise program for individuals with COPD and compare the outcomes with those achieved through standard care.

Individuals with COPD who have completed a previous rehabilitation program will be enrolled in the study. Study participants will be assigned randomly to either a year-long community exercise program or usual care. Those assigned to the community program will exercise twice weekly at a local community centre supervised by trained fitness instructors. A case manager will facilitate the transition from the hospital rehabilitation program to the community centre. The case manager will also be available to participants and instructors for consult as needed. Continuing to build on an established partnership with the City of Toronto, the case manager will ensure fitness instructors receive specialized training in order to properly supervise and support the individuals with COPD. Participants assigned to usual care group will receive standard care by their family physician and respiratory specialist. Functional status will be evaluated before the program begins and again at 6-months and 1-year. The outcome of each group will be compared to determine the effectiveness of the community exercise program. It is hypothesized that individuals who participate in the community exercise program will have better function and quality of life versus those individuals who receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* individuals with moderate to severe COPD based on international (GOLD) criteria
* clinically stable
* able to provide their own informed consent
* able to secure independent transportation to the community site

Exclusion Criteria:

* individuals with associated medical conditions that limit their exercise tolerance (cardiovascular, musculo-skeletal, recent surgery, etc.)
* individuals who report a history of significant cardiovascular disease (i.e. congestive cardiac failure, history of cardiac arrest, acute myocardial infarction within the preceding three months, symptomatic ischaemic cardiac disease, uncontrolled systemic hypertension) or report severe non-respiratory symptoms during exercise
* individuals receiving mechanical ventilation
* individuals who are unable to attend the community-based exercise program or follow-up assessment sessions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-11; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Six Minute Walk Test at 6 months | Baseline and 6 months
Change from baseline in Six Minute Walk Test at 12 months | Baseline and 12 months

SECONDARY OUTCOMES:
Change from baseline in Chronic Respiratory Disease Questionnaire at 6 months | Baseline and 6 months
Change from baseline in Repeated Chair Stand at 6 months | Baseline and 6 months
Change from baseline in Duke Activity Status Index at 6 months | Baseline and 6 months
Change from baseline in Health Utilities Index at 6 months | Baseline and 6 months
Change in baseline in COPD Self-Efficacy Scale at 6 months | Baseline and 6 months
Change from baseline in Chronic Respiratory Disease Questionnaire at 12 months | Baseline and 12 months
Change from baseline in Duke Activity Status Index at 12 months | Baseline and 12 months
Change from baseline in Health Utilities Index at 12 months | Baseline and 12 months
Change from baseline in Repeated Chair Stand at 12 months | Baseline and 12 months
Change in baseline in COPD Self-Efficacy Scale at 12 months | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, MD, Principal Investigator — West Park Healthcare Centre
Locations (4):
- Canada (4):
  - Trillium Health Partners- Credit Valley Hospital, Mississauga, Ontario
  - St. Joseph's Care Group, Thunder Bay, Ontario
  - West Park Healthcare Centre, Toronto, Ontario
  - Lakeridge Health, Whitby, Ontario